CLINICAL TRIAL: NCT02920151
Title: Effects of Balance Exercises Circuit in Patients With Total Hip or Knee Arthroplasty (BECA): A Randomized Clinical Trial
Brief Title: Effects of Balance Exercises Circuit in Patients With Hip or Knee Arthroplasty
Acronym: BECA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo de Estudos e Pesquisas Sobre Atividade Física Para Idosos (Other)
Responsible Party: Principal Investigator, Marisete Peralta Safons, professor, Grupo de Estudos e Pesquisas Sobre Atividade Física Para Idosos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Gepafi
Record Dates: First submitted 2016-09-12; First posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Hip Replacement; Knee Replacement; Postural Balance
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BALANCE EXERCISES CIRCUIT (Experimental): balance exercises circuit for three months, twice weekly, 50 minutes per day.
  Interventions: Other: balance exercises circuit
- CONTROL GROUP (No Intervention): usual routine

INTERVENTIONS:
Other: balance exercises circuit — Thirteen workstations were organized in a circuit format on involved multidirectional gait in different bases of support, unstable surfaces, functional reach, exercise with balls, and single-leg stance
  Other Names: exercises
  Arms: BALANCE EXERCISES CIRCUIT

SUMMARY:
This study evaluates the effect of balance circuit in patients with more than one year of postoperative total hip or knee arthroplasty. Patients were randomized between intervention group (IG) (balance exercise circuit ) and control group (CG) (usual routine). The evaluations were conducted by blind examiners.

DETAILED DESCRIPTION:
Balance Exercise Circuit (BEC) program, includes exercise that specifically challenge sensory inputs from mechanoreceptors as well as from the visual and vestibular systems. It is composed of 13 stations, involving static and dynamic balance exercises, including tandem walking, forward-backward stepping, wide-stance gait, functional reach, heel lift, toe press, balance on unstable surfaces, and standing on one leg. The BEC lasts 50 min, two times per week for a total of 12 weeks. Progression of exercises occurred every 3 weeks and was closely supervised to ensure safety. Each BEC session comprised of warm-up and stretching (10 min), exercise circuit (30 min), and cool-down (10 min).

ELIGIBILITY:
Inclusion Criteria:

* more than one year of postoperative total hip or knee arthroplasty

Exclusion Criteria:

* total hip AND knee arthroplasty
* other surgeries of the lower limbs and spine
* autoimmune disease
* contraindication for physical exercise

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | three months
  evaluates functional balance

SECONDARY OUTCOMES:
QuickScreen scale | three months
  fall risk assessement
Falls Efficacy Scale | three months
  self-efficacy or confidence in performing activities without falling

OTHER OUTCOMES:
static balance | three months
  static balance assessed by force plate
Timed Up and Go | three months
  functional performance and functional balance

CONTACTS AND LOCATIONS:
Overall Officials: Marisete P Safons, Principal Investigator — Grupo de Estudos e Pesquisas Sobre Atividade Física Para Idosos

IPD SHARING:
Plan to Share IPD: No